CLINICAL TRIAL: NCT06752356
Title: A Double-blind, Randomized, Multi-Center Study Investigating Efficacy and Safety of Two Different Dosages of Intravenous Human Normal Immune Globulin (IGIV) 10% in Subjects With Chronic Inflammatory Demyelinating Polyneuropathy (CIDP)
Brief Title: A Study Investigating Intravenous Human Normal Immune Globulin (IGIV) 10% in Subjects With Chronic Inflammatory Demyelinating Polyneuropathy (CIDP)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kedrion S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-518596-61-00; KB071 (Other: Kedrion S.p.A)
Record Dates: First submitted 2024-12-16; First posted 2024-12-30 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy
Keywords: Chronic Inflammatory Demyelinating Polyneuropathy; CIDP; Intravenous; Human Immunoglobulin; KIg10
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — Immunoglobulins; Solutions; Administration, Intravenous

STUDY DESIGN:
Intervention Model Description: Double Blind, Randomized.
Who Masked: Participant, Investigator
Masking Description: Sponsor will also be masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1.0 g/kg dose group for 24 weeks (Experimental): This group will receive, initial loading dose of 2.0 g/kg of Intravenous (IV) KIg10 (Immunoglobulin) infusion followed by 1.0 g/kg of IV KIg10 every 3 weeks.
  Interventions: Biological: Immune globulin (human) 10% solution for intravenous administration
- 0.5 g/kg dose group for 24 weeks (Experimental): This group will receive, Initial loading dose of 2.0 g/kg of Intravenous (IV) KIg10 (Immunoglobulin) infusion will be given followed by 0.5 g/kg of IV KIg10 every 3 weeks.
  Interventions: Biological: Immune globulin (human) 10% solution for intravenous administration

INTERVENTIONS:
Biological: Immune globulin (human) 10% solution for intravenous administration — Kedrion intravenous immunoglobulin (IVIg) 10%
  Other Names: KIg10

SUMMARY:
The current study is being conducted to assess the efficacy and safety of KIg10 (Intravenous Human Immune globulin 10%) at two different dosages as maintenance therapy for Chronic Inflammatory Demyelinating Polyneuropathy (CIDP) following 21 weeks of treatment.

DETAILED DESCRIPTION:
This is a Double Blind, Randomized study. All subjects will enter a wash-out phase of up to 12 weeks, or until functional deterioration, defined as an increase of ≥1 point (worsening) in the adjusted INCAT disability score, is demonstrated. Eligible subjects will then be randomized in a 1:2 ratio to receive either 0.5 g/kg or 1.0 g/kg KIg10 at 3-weekly intervals for 21 weeks. Subjects who relapse during randomized treatment due to functional deterioration, based on the INCAT score, will be rescued with 2.0 g/kg KIg10 at 3-weekly intervals for 21 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥18 years.
2. Written informed consent and authorization to access personal health information obtained independently from subjects indicating that they understand the purpose of, and procedures required for, the study and are willing to participate.
3. Documented diagnosis of chronic inflammatory demyelinating polyradiculoneuropathy (CIDP) consistent with the 2021 EAN/PNS criteria.
4. Current or documented history of significant disability, as defined by an overall adjusted INCAT disability score between 2 and 9. A score of 2 must be exclusively from the lower extremities.
5. Subjects are currently dependent on treatment with immunoglobulins, corticosteroids, or standard of care treatments for CIDP.
6. Weakness of at least two limbs.
7. Subjects should be clinically stable 12 weeks prior to screening date as defined by:

   * without a worsening in INCAT score of ≥1 point, AND/OR
   * without significant changes in clinical symptoms, AND
   * without significant dose changes or requiring additional treatments.

Exclusion Criteria:

1. Pure sensory atypical and multivariant CIDP.
2. Females who are pregnant, breastfeeding, unwilling to practice adequate contraception throughout the study or planning a pregnancy during the course of the study.
3. IG-experienced subjects requiring an IGIV dosage of more than 1.3 g/kg/month OR SCIG pre-treated subjects requiring a SCIG dosage of more than 1.6 g/kg/month.
4. Subjects who have previously failed to respond to IGIV or SCIG.
5. On screening date, a body mass index (BMI) > 35 kg/m2 or an IGIV dose that puts the patient at risk of fluid overload.
6. CIDP and any neuropathy of other causes not consistent with the 2021 EAN/PNS criteria.
7. Immunoglobulin M (IgM) paraproteinemia, including IgM monoclonal gammopathy with high titer antibodies to myelin-associated glycoprotein.
8. Central demyelinating disorders (e.g, multiple sclerosis) or severe myopathy.
9. Any chronic or debilitating disease, or central nervous disorder that causes neurological symptoms or may interfere with assessment of CIDP or outcome measures
10. Congestive heart failure (New York Heart Association (NYHA) Class III/IV), unstable angina, unstable cardiac arrhythmias, or uncontrolled hypertension
11. History of deep vein thrombosis or thromboembolic events (e.g, cerebrovascular accident, pulmonary embolism) in the past 12 months.
12. Condition(s) which could alter protein catabolism and/or IgG utilization (e.g, protein-losing enteropathies, nephrotic syndrome).
13. Known history of chronic kidney disease, or glomerular filtration rate (GFR) of <60 milliliter per minute per 1.73 square meter (mL/min/1.73m2) estimated based on an established CKD-EPI equation at the time of screening.
14. Active malignancy requiring chemotherapy and/or radiotherapy, or history of malignancy with less than 2 years of complete remission prior to screening. Exceptions are: adequately treated basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, and stable prostate cancer not requiring treatment.
15. Hypersensitivity or adverse reactions (e.g, urticaria, breathing difficulty, severe hypotension, or anaphylaxis) to human blood products such as human IgG, albumin, or other blood components.
16. Known history of immunoglobulin A (IgA) deficiency.
17. Known history of autoimmune nodo-paranodopathies causing IG treatment resistance.
18. Abnormal laboratory values at screening:

    1. Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) > 2.5x upper limit of normal (ULN)
    2. Platelet count <100,000 cells/µL.
    3. Absolute neutrophil count (ANC) <1000 cells/µL.
    4. Clinically significant anemia defined as hemoglobin (Hgb) level of < 10.0 g/dL at screening.
19. Ongoing/active infection with hepatitis B virus (HBV), hepatitis C virus (HCV) or HIV Type 1/2 infection. Subjects with chronic hepatitis B or hepatitis C infection currently on treatment may participate as long as they have undetectable viral load within 12 months of screening date.
20. Subjects who have received:

    1. Within 2 months before wash-out phase:

       * plasma exchange
       * change in treatment of methotrexate, azathioprine, or mycophenolate
    2. Within 3 months before wash-out phase: Efgartigimod alfa (Vyvgart)
    3. Within 5 months before wash-out phase: cyclophosphamide, interferon, tumor necrosis factor-alpha inhibitors, fingolimod, or any other immunosuppressive medications
    4. Within 12 months before wash-out phase: rituximab or alemtuzumab
21. Subjects who have received a hematopoietic stem cell transplant.
22. Subjects on corticosteroids for the treatment of CIDP after being fully washed out. Subjects on maintenance doses of corticosteroid may be allowed, if treatment is for conditions unrelated to CIDP (doses usually below 20 mg/day prednisone or equivalent and where the dosage is unlikely to be tapered during the duration of the trial may be allowed).
23. Any disorder or condition that in the investigator's judgment may impede the subject's participation in the study, pose increased risk to the subject, or confound the results of the study.
24. Participation in another clinical study involving an investigational product (IP) or investigational device within 30 days prior to screening visit or is scheduled to participate in another clinical study involving an IP or investigational device during the intended course of this study.
25. History of acquired or inherited thrombophilic disorders. These will include the specific types of acquired or inherited thrombophilic disorders that could put subjects at risk of developing thrombotic events.
26. Previous participation in this clinical study.
27. Any other factor that, in the opinion of the investigator, would prevent the subject from complying with the requirements of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12-20 (Estimated); Study Completion 2027-12-27 (Estimated)

PRIMARY OUTCOMES:
Efficacy of 1.0 g/kg KIg10 in the treatment of adult subjects with active CIDP | From Baseline upto 24 weeks of treatment
  The proportion of responders in the 1.0 g/kg KIg10 arm, at week 24 relative to Randomization Baseline week 0, based on the adjusted INCAT disability score. A responder is defined as having a ≥1 point decrease (improvement) in the adjusted INCAT score at week 24 relative to adjusted INCAT score at randomization baseline.

SECONDARY OUTCOMES:
Efficacy of 0.5 g/kg KIg10 in the treatment of adult subjects with active CIDP | From Baseline upto 24 weeks of treatment
  The proportion of responders in the 0.5 g/kg KIg10 arm at week 24 relative to randomization baseline, based on the adjusted INCAT disability score. A responder is defined as having a ≥1 point decrease (improvement) in the adjusted INCAT score at week 24 relative to adjusted INCAT score at randomization baseline.
Proportion of responders (Week 24 vs Baseline) in both dose groups | From Baseline upto 24 weeks of treatment
  Proportion of responders in both dose groups based on Grip Strength and I-RODs
Proportion of responders in rescued subjects | End of Treatment vs onset of rescue treatment
  Proportion of responders in rescued subjects based on grip strength, I-RODS scores, adjusted INCAT disability score
Improvers based on the MRC-sumscore | From Baseline upto 24 weeks of treatment
  Improvers by a change of 4 points in both dose groups (week 24 versus baseline) based on MRC-sumscore
Mean Change in MRC-sumscore | From Baseline upto 24 weeks of treatment
  Mean change in MRC-sumscore for both dose groups at week 24 vs baseline
Mean Change in MRC-sumscore for rescued subjects | End of Treatment vs onset of rescue treatment
  Mean change in MRC-sumscore for rescued subjects from End of Treatment versus onset of rescue treatment
Disease Related QoL (CAPPRI) for each dose level | From Baseline upto 24 weeks of treatment
  For each dose level the Chronic Acquired Polyneuropathy Patient Reported Index (CAPPRI) will be analysed for disease related QoL
Mean change in I-RODS | From Baseline upto 24 weeks of treatment
  For each dose level, mean change from randomization baseline (visit 2, week 0) to end of study (visit 10, week 24) in Inflammatory-Rasch-built Overall Disability Scale (I- RODS) score
Mean change in I-RODS for rescued subjects | End of Treatment vs onset of rescue treatment
  Mean change to the end of treatment assessments prior to onset of rescue treatment, in Inflammatory-Rasch-built Overall Disability Scale (I- RODS) score for rescued subjects

OTHER OUTCOMES:
Number of adverse events | From Baseline upto 25 weeks
  Assess Safety and Tolerability of KIg10
The proportion of patients experiencing at least one adverse event. | From Baseline upto 25 weeks
  Assess Safety and Tolerability of KIg10

CONTACTS AND LOCATIONS:
Overall Officials: Miranda Norton, PhD, Study Chair — Kedrion S.p.A.
Locations (1):
- Advanced Neurology Epilepsy and Sleep Center/ANESC Research, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR

REFERENCES:
- [Background] Hughes RA, Donofrio P, Bril V, Dalakas MC, Deng C, Hanna K, Hartung HP, Latov N, Merkies IS, van Doorn PA; ICE Study Group. Intravenous immune globulin (10% caprylate-chromatography purified) for the treatment of chronic inflammatory demyelinating polyradiculoneuropathy (ICE study): a randomised placebo-controlled trial. Lancet Neurol. 2008 Feb;7(2):136-44. doi: 10.1016/S1474-4422(07)70329-0. PMID 18178525
- See also: Lewis et al. Chronic Inflammatory Demyelinating Polyneuropathy, National Organization for Rare Disorders, Updated 01Oct2024 — https://rarediseases.org/rare-diseases/chronic-inflammatory-demyelinating-polyneuropathy/